CLINICAL TRIAL: NCT04072484
Title: Effectiveness of Chest Compressions Under Mild Hypoxia: Should Rescuers Breathe Supplemental Oxygen on Commercial Flights?
Brief Title: Effectiveness of Chest Compressions Under Mild Hypoxia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research at the University of Chicago was halted in March 2020.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB19-0535
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Arrest; Hypoxia
MeSH Terms: conditions — Heart Arrest; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant is unaware of the oxygen concentration that he or she is breathing during either arm of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Room Air (No Intervention): The reduced oxygen breathing device will be set to deliver room air. (i.e., no oxygen is removed from the gas mixture. The subject will perform CPR while breathing through mask and tubing that is connected to the device.
- Hypoxia (Experimental): The reduced oxygen breathing device will be set to deliver a gas mixture with15% oxygen. (Equivalent to the partial pressure of oxygen at 2,438 meters.) The subject will perform CPR while breathing through mask and tubing that is connected to the device.
  Interventions: Other: Mild hypoxia

INTERVENTIONS:
Other: Mild hypoxia — The subject will breathe a gas mixture containing 15% oxygen instead of 21% oxygen.
  Arms: Hypoxia

SUMMARY:
The purpose of this study is to evaluate the effect of breathing a slightly reduced amount of oxygen will have on a rescuer's ability to provide chest compressions during CPR.

DETAILED DESCRIPTION:
Cardiac arrest can occur in any setting, even flying on a commercial airliner, and chest compressions are a critical, lifesaving component of cardiopulmonary resuscitation (CPR). If a cardiac arrest occurs on board a commercial flight, CPR may be administered by cabin crew members or health care professionals who are passengers and volunteer their assistance. The in-flight environment presents significant challenges, including an unfamiliar environment, an unknown patient, cramped space, and the fact that the pressure altitude in the cabin is between 6,000 feet and 8,000 feet. Even though the fraction of inspired oxygen (FiO2) is still 0.21, with decreased pressure the rescuer is effectively breathing a FiO2 of 0.15 and is mildly hypoxic. Although the decreased PaO2 seen in even in healthy passengers is a normal occurrence when flying on a commercial airliner, it may impair the ability of a rescuer to perform adequate CPR. Administering supplemental oxygen to the rescuer may enable provision of more effective chest compressions. In this study, we will measure the quality of chest compressions in normoxic and hypoxic conditions during short simulation scenarios. We hypothesize that chest compressions will be more effective in a normoxic environment.

All tasks are being performed for research purposes. All tasks will take place at the University of Chicago in an empty conference room. After the pre-study screening survey, subjects will be asked to perform chest compressions during a simulated cardiac arrest and will then fill out a survey. Subjects will participate in 2 sessions each; the sessions will be at least one day apart. During each session, the subject will wear a face mask. Subjects will be randomized and blinded to one of two conditions: During CPR, the subject will receive a FiO2 of 0.21 or 0.15 by face mask, which will produce a partial pressure of oxygen similar to, but slightly higher than, that of a commercial airliner. The gas mixture will be delivered by a normobaric hypoxia training device. During the second session, subjects will receive the other oxygen concentration.

Each session will consist of a simulation in which a passenger on an airplane (i.e., a mannequin) has an asystolic cardiac arrest. Participants will provide compression-only CPR. Every 2 minutes, the preceptor will ask the subject stop compressions for 10 seconds for a pulse and rhythm check, similar to actual established protocols. The participant will be wearing a pulse oximeter. The scenario will end after 30 minutes (14 rounds of 2 minutes each of CPR by the subject, consistent with the Universal Guidelines for Termination of CPR), or if the subject becomes fatigued and wishes to stop or is no longer providing high quality chest compressions.

ELIGIBILITY:
Inclusion Criteria:

* Previous CPR training
* Baseline exercise tolerance of at least 4 metabolic equivalents (METS)

Exclusion Criteria:

* Heart disease
* Moderate or severe asthma
* Carpal tunnel syndrome
* Mononucleosis
* Respiratory infections
* Current injury (e.g., sprain, fracture, or dislocation)
* Acute or chronic muscle or joint pain
* Recent exposure to high altitude
* Any other condition that limits physical activity
* Any condition that precludes flying on a commercial airline flight

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Successful CPR | 30 minutes
  Number of successful two-minute CPR rounds

SECONDARY OUTCOMES:
Lowest oxygen saturation | 30 minutes
  Lowest oxygen saturation observed during CPR
Survey results - Fatigue | 30 minutes
  Participants will rate their level of fatigue on a scale from 0 - 100 (100 = maximum fatigue)
Survey results - Chest compression | 30 minutes
  Participants will rate the quality of chest compressions on a scale from 0 - 100 (100 = best chest compressions)

CONTACTS AND LOCATIONS:
Overall Officials: Keith J Ruskin, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleinman ME, Goldberger ZD, Rea T, Swor RA, Bobrow BJ, Brennan EE, Terry M, Hemphill R, Gazmuri RJ, Hazinski MF, Travers AH. 2017 American Heart Association Focused Update on Adult Basic Life Support and Cardiopulmonary Resuscitation Quality: An Update to the American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2018 Jan 2;137(1):e7-e13. doi: 10.1161/CIR.0000000000000539. Epub 2017 Nov 6. PMID 29114008
- [Background] Ruskin KJ, Ricaurte EM, Alves PM. Medical Guidelines for Airline Travel: Management of In-Flight Cardiac Arrest. Aerosp Med Hum Perform. 2018 Aug 1;89(8):754-759. doi: 10.3357/AMHP.5038.2018. PMID 30020062
- [Background] Muhm JM. Predicted arterial oxygenation at commercial aircraft cabin altitudes. Aviat Space Environ Med. 2004 Oct;75(10):905-12. PMID 15497372
- [Background] Kwak SJ, Kim YM, Baek HJ, Kim SH, Yim HW. Chest compression quality, exercise intensity, and energy expenditure during cardiopulmonary resuscitation using compression-to-ventilation ratios of 15:1 or 30:2 or chest compression only: a randomized, crossover manikin study. Clin Exp Emerg Med. 2016 Sep 30;3(3):148-157. doi: 10.15441/ceem.15.105. eCollection 2016 Sep. PMID 27752633
- [Background] Romer LM, Haverkamp HC, Amann M, Lovering AT, Pegelow DF, Dempsey JA. Effect of acute severe hypoxia on peripheral fatigue and endurance capacity in healthy humans. Am J Physiol Regul Integr Comp Physiol. 2007 Jan;292(1):R598-606. doi: 10.1152/ajpregu.00269.2006. Epub 2006 Sep 7. PMID 16959862
- [Background] Drennan IR, Case E, Verbeek PR, Reynolds JC, Goldberger ZD, Jasti J, Charleston M, Herren H, Idris AH, Leslie PR, Austin MA, Xiong Y, Schmicker RH, Morrison LJ; Resuscitation Outcomes Consortium Investigators. A comparison of the universal TOR Guideline to the absence of prehospital ROSC and duration of resuscitation in predicting futility from out-of-hospital cardiac arrest. Resuscitation. 2017 Feb;111:96-102. doi: 10.1016/j.resuscitation.2016.11.021. Epub 2016 Dec 5. PMID 27923115
- [Background] Wang JC, Tsai SH, Chen YL, Hsu CW, Lai KC, Liao WI, Li LY, Kao WF, Fan JS, Chen YH. The physiological effects and quality of chest compressions during CPR at sea level and high altitude. Am J Emerg Med. 2014 Oct;32(10):1183-8. doi: 10.1016/j.ajem.2014.07.007. Epub 2014 Jul 30. PMID 25154345